CLINICAL TRIAL: NCT00510627
Title: A Prospective, Randomized, Active-Control, Multi-Center Study Assessing Overall Survival Using Chemotherapy With or Without Impedance-Based Radiofrequency Ablation for Subjects With Colorectal Cancer and Incurable Metastatic Liver Disease, Failing at Least First-Line Chemotherapy
Brief Title: Study Comparing Radio Frequency Ablation Plus Chemotherapy and Chemotherapy Alone in Patients With Secondary Liver Metastases
Acronym: Prometheus
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Boston Scientific has decided to close the Study.
Sponsor: Boston Scientific Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONC-PM-032006
Record Dates: First submitted 2007-07-31; First posted 2007-08-02 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Metastatic Liver Cancer; Secondary Liver Cancer; Liver Neoplasm
Keywords: Metastatic Liver Cancer; Colorectal Cancer; Radiofrequency Ablation; Chemotherapy
MeSH Terms: conditions — Liver Neoplasms; Colorectal Neoplasms | interventions — Radiofrequency Ablation; Radionuclide Generators; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Radiofrequency ablation in conjunction with chemotherapy
  Interventions: Device: Radiofrequency Ablation (RFA)
- B (Active Comparator): Standard of care chemotherapy regimen
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Device: Radiofrequency Ablation (RFA) — The RF3000 radiofrequency generator has the capacity to deliver 200 watts of alternating current to the needle electrode for the coagulation necrosis of soft tissue.
  Other Names: RF3000 Radiofrequency (RF) Generators; LeVeen Electrode; Co-Access Electrode; Soloist Electrode; SuperSlim Electrode
  Arms: A
Drug: Chemotherapy — Standard of care chemotherapy regimen
  Other Names: Oxaliplatin containing chemotherapy regimen; Irinotecan containing chemotherapy regimen; An anti-EGFR monoclonal antibody-containing regimen; Other
  Arms: B

SUMMARY:
The purpose of this study is to determine whether patients treated with Radiofrequency Ablation (RFA) in conjunction with chemotherapy have a better overall survival rate than patients treated with chemotherapy alone.

DETAILED DESCRIPTION:
The American Cancer Society has estimated that colorectal cancer is the second leading cause of cancer related deaths, with 106,370 new cases diagnosed in 2004. Due to the unique nature of the hepatic circulatory system, with preferential portal venous drainage of the gastrointestinal tract, the liver is the most common site for metastatic tumor growth from a colorectal carcinoma. It is estimated that approximately 20% of patients diagnosed with colorectal cancer will present with liver involvement at the time of diagnosis, and 50% of patients will manifest metastatic involvement of the liver following resection of the primary colorectal cancer. Over one half of patients who die of colorectal cancer have liver metastases at autopsy.

The current "gold standard" in the treatment of isolated metastatic liver disease is curative hepatic resection. Only within the last 20 years has surgical resection become a viable option, as in the past it was considered unjustified due to high morbidity and mortality rates. The primary drawback to hepatic resection is the sheer number of patients for whom it is contraindicated. Only 10-20% of patients liver metastases are candidates for surgical resection, owing to factors such as tumor locations, size, extent of disease, and other medical co-morbidities.

Historically, in cases where hepatic resection was contraindicated, systemic chemotherapy was the only alternative treatment. In the last several years an increasing number of hepatic directed therapies have become available such as hepatic artery ligation, radiation, hepatic artery infusion of chemotherapy, chemoembolization, and mechanical ablation of the tumor(s).

One mechanical method of ablation involves the use of radiofrequency thermal technology, also called radiofrequency ablation (RFA). The RFA procedure involves inserting an RF electrode into the center of a hepatic tumor mass under ultrasonic or CT guidance. Radiofrequency energy is then applied through the electrode, causing a thermal injury to the surrounding tumor tissue. Currently there are two basic designs for monitoring inter-procedural progress during RFA; temperature monitoring of set points within the target tissue with thermocouples, or assessing the system-wide impedance of tissue adjacent to the deployed electrode tines. Radiofrequency ablation systems are comprised of three components: a radiofrequency generator, an active electrode, and dispersive electrodes.

To date no prospective multi-center trials have been completed which would conclusively demonstrate whether RFA is an effective adjunct to systemic chemotherapy with respect to advantages in median overall survival compared with chemotherapy alone. The primary objective of this trial is to determine overall survival for subjects with colorectal cancer and incurable metastatic liver disease who fail at least first line chemotherapy and are treated with radiofrequency ablation plus additional chemotherapy, compared to subjects receiving additional chemotherapy only.

ELIGIBILITY:
Inclusion Criteria:

All subjects must meet the following criteria:

* Subject must have incurable metastatic colorectal cancer with metastatic disease to the liver
* Subject must have extrahepatic metastatic disease, as confirmed by radiographic evidence or surgical/other documentation that cannot be treated by surgery or image guided therapy to an endpoint of no evidence of residual disease by imaging criteria
* Subject has received and, in the opinion of the treating physician, progressed through at least one prior chemotherapy regimen for metastatic disease, or has developed recurrent disease on or within 6 months of completing adjuvant therapy
* At least 50% of the total tumor burden is in the liver, as determined by the treating investigator, and prior to any study specified intervention (resection or ablation).
* Subject must have no more than 10 hepatic tumors remaining after surgical resection, with no tumor exhibiting a unidimensional size greater than 5cm
* Subject is medically eligible to receive RFA, as determined by the treating investigator
* Subject is naïve to, and medically eligible (as defined by the treating investigator) to receive, at least one of the following:
* an oxaliplatin containing regimen
* an irinotecan containing regimen
* an anti-EGFR monoclonal antibody-containing regimen (subject must be naïve to both cetuximab and panitumumab)
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
* Age > 18 years
* Subject life expectancy > 3 months
* International Normalized Ratio (INR) < 2.0
* Platelets > 100 x103/mm3
* Total Bilirubin <1.5mg/dl
* Creatinine level < 2.0 mg/dl
* Must sign an Informed Consent form

Exclusion Criteria:

All subjects who meet any of the following criteria will not be enrolled into the study:

* Subjects's extrahepatic disease is amenable to curative surgical or image guided therapy
* Subject has known brain metastases
* Uncorrectable coagulopathy
* Subject is pregnant, nursing, or wishes to become pregnant during the study
* Other serious medical condition(s) (e.g. uncontrolled infection, uncontrolled cardiac disease) that, in the opinion of the treating investigator, would preclude study treatment or impact survival.
* Current or planned treatment with any experimental chemotherapy or biological agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-08; Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate Overall Survival in subjects receiving chemotherapy + RFA compared to chemotherapy alone. | Study duration

SECONDARY OUTCOMES:
To evaluate any unanticipated adverse device effects. | Two years
To determine if there are differences in the incidence or severity of adverse events in the RFA + chemotherapy arm compared to the chemotherapy only arm. | Study duration

CONTACTS AND LOCATIONS:
Overall Officials: William Jacqmein, Study Director — Boston Scientific Corporation
Locations (2):
- United States (2):
  - New York University, New York, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio

REFERENCES:
- [Background] Chapter 49, Colon, Rectal, and Anal Cancers. PART VI: THE CARE OF INDIVIDUALS WITH SPECIFIC CANCERS; pp: 1156-1214
- [Background] Choti MA, Bulkley GB. Management of hepatic metastases. Liver Transpl Surg. 1999 Jan;5(1):65-80. doi: 10.1002/lt.500050113. PMID 9873095
- [Background] Cromheecke M, de Jong KP, Hoekstra HJ. Current treatment for colorectal cancer metastatic to the liver. Eur J Surg Oncol. 1999 Oct;25(5):451-63. doi: 10.1053/ejso.1999.0679. PMID 10527592
- [Background] Kemeny NE, Atiq OT. Non-surgical treatment for liver metastases. Baillieres Best Pract Res Clin Gastroenterol. 1999 Dec;13(4):593-610. doi: 10.1053/bega.1999.0050. PMID 10654922
- [Background] Fong Y. Surgical therapy of hepatic colorectal metastasis. CA Cancer J Clin. 1999 Jul-Aug;49(4):231-55. doi: 10.3322/canjclin.49.4.231. PMID 11198884
- [Background] Bowles BJ, Machi J, Limm WM, Severino R, Oishi AJ, Furumoto NL, Wong LL, Oishi RH. Safety and efficacy of radiofrequency thermal ablation in advanced liver tumors. Arch Surg. 2001 Aug;136(8):864-9. doi: 10.1001/archsurg.136.8.864. PMID 11485520
- [Background] Berber E, Pelley R, Siperstein AE. Predictors of survival after radiofrequency thermal ablation of colorectal cancer metastases to the liver: a prospective study. J Clin Oncol. 2005 Mar 1;23(7):1358-64. doi: 10.1200/JCO.2005.12.039. Epub 2005 Jan 31. PMID 15684312
- [Background] Yoon SS, Tanabe KK. Surgical treatment and other regional treatments for colorectal cancer liver metastases. Oncologist. 1999;4(3):197-208. PMID 10394588
- [Background] DeMatteo RP, Fong Y, Blumgart LH. Surgical treatment of malignant liver tumours. Baillieres Best Pract Res Clin Gastroenterol. 1999 Dec;13(4):557-74. doi: 10.1053/bega.1999.0048. PMID 10654920
- [Background] Curley SA, Vecchio R. New trends in the surgical treatment of colorectal cancer liver metastases. Tumori. 1998 May-Jun;84(3):281-8. doi: 10.1177/030089169808400301. PMID 9678609
- [Background] Dodd GD 3rd, Soulen MC, Kane RA, Livraghi T, Lees WR, Yamashita Y, Gillams AR, Karahan OI, Rhim H. Minimally invasive treatment of malignant hepatic tumors: at the threshold of a major breakthrough. Radiographics. 2000 Jan-Feb;20(1):9-27. doi: 10.1148/radiographics.20.1.g00ja019. PMID 10682768
- [Background] Poston GJ. Radiofrequency ablation of colorectal liver metastases: where are we really going? J Clin Oncol. 2005 Mar 1;23(7):1342-4. doi: 10.1200/JCO.2005.10.911. Epub 2005 Jan 31. No abstract available. PMID 15684315
- [Background] Pawlik TM, Abdalla EK, Ellis LM, Vauthey JN, Curley SA. Debunking dogma: surgery for four or more colorectal liver metastases is justified. J Gastrointest Surg. 2006 Feb;10(2):240-8. doi: 10.1016/j.gassur.2005.07.027. PMID 16455457
- [Background] Tournigand C, Andre T, Achille E, Lledo G, Flesh M, Mery-Mignard D, Quinaux E, Couteau C, Buyse M, Ganem G, Landi B, Colin P, Louvet C, de Gramont A. FOLFIRI followed by FOLFOX6 or the reverse sequence in advanced colorectal cancer: a randomized GERCOR study. J Clin Oncol. 2004 Jan 15;22(2):229-37. doi: 10.1200/JCO.2004.05.113. Epub 2003 Dec 2. PMID 14657227
- [Background] Giantonio et. Al. High-dose bevacizumab in combination with FOLFOX4 improves survival in patients with previously treated advanced colorectal cancer: Results from the Eastern Cooperative Oncology Group (ECOG) study E3200
- [Background] Talamonti MS, Tellez C, Benson AB 3rd. Local-regional therapy for metastatic liver tumors. Cancer Treat Res. 1998;98:172-99. No abstract available. PMID 10326669